CLINICAL TRIAL: NCT02491333
Title: The Effect of Acupuncture on Insulin Sensitivity of Women With Polycystic Ovary Syndrome and Insulin Resistance: a Randomized Controlled Trial
Brief Title: The RCT of Acupuncture on PCOS Combined With IR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: The University of Hong Kong (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Hongxia Ma, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCOSIRct
Record Dates: First submitted 2015-06-24; First posted 2015-07-08 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
Keywords: polycystic ovary syndrome; acupuncture; insulin resistance; HOMA-IR; metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- true acupuncture + placebo metformin (Experimental): True acupuncture and placebo metformin will be started 2 days after the baseline visit including OGTT. All subjects will be asked to use a barrier method for contraception.
  True acupuncture treatment will be given three times per week. Each treatment session lasts for 30 minutes and can be separated by an interval of 1-3 days, with a maximum of 48 treatment sessions during 4 month.
  Placebo metformin will be given at 0.5g/times, 3 times one day and for 4 month.
  Interventions: Other: true acupuncture; Drug: Placebo metformin
- sham acupuncture + placebo metformin (Sham Comparator): Sham acupuncture and placebo metformin will be started 2 days after the baseline visit including OGTT. All subjects will be asked to use a barrier method for contraception.
  Sham acupuncture treatment will be given three times per week. Each treatment session lasts for 30 minutes and can be separated by an interval of 1-3 days, with a maximum of 48 treatment sessions during 4 month. Placement of needles is unlikely to affect ovulation and IR in women with PCOS.
  Placebo metformin will be given at 0.5g/times, 3 times one day and for 4 month.
  Interventions: Other: sham acupuncture; Drug: Placebo metformin
- sham acupuncture + metformin (Active Comparator): Sham acupuncture and metformin will be started 2 days after the baseline visit including OGTT. All subjects will be asked to use a barrier method for contraception.
  Sham acupuncture treatment will be given three times per week. Each treatment session lasts for 30 minutes and can be separated by an interval of 1-3 days, with a maximum of 48 treatment sessions during 4 month.Placement of needles is unlikely to affect ovulation and IR in women with PCOS.
  Metformin will be given at 0.5g/times, 3 times one day and for 4 month.
  Interventions: Other: sham acupuncture; Drug: metformin

INTERVENTIONS:
Other: true acupuncture — True acupuncture treatment will be given three times per week. Each treatment session lasts for 30 minutes and can be separated by an interval of 1-3 days, with a maximum of 48 treatment sessions during 4 month.
  Arms: true acupuncture + placebo metformin
Other: sham acupuncture — Sham acupuncture treatment will be given three times per week. Each treatment session lasts for 30 minutes and can be separated by an interval of 1-3 days, with a maximum of 48 treatment sessions during 4 month.
  Arms: sham acupuncture + metformin; sham acupuncture + placebo metformin
Drug: metformin — Metformin will be given at 0.5g/times, 3 times one day and for 4 month.
  Other Names: Dimethylbiguanide
  Arms: sham acupuncture + metformin
Drug: Placebo metformin — Placebo metformin will be given at 0.5g/times, 3 times one day and for 4 month.
  Other Names: placebo Dimethylbiguanide
  Arms: sham acupuncture + placebo metformin; true acupuncture + placebo metformin

SUMMARY:
The objectives of this randomized controlled trial are to compare insulin sensitivity following true acupuncture + placebo metformin (Group 1) vs sham acupuncture + placebo metformin (Group 2) vs sham acupuncture + metformin (Group 3) in women with PCOS and IR.

DETAILED DESCRIPTION:
1.1 Study design This is a randomized double blind controlled. 1.2 Subject selection and exclusion Women with PCOS and IR will be recruited from the Department of Traditional Chinese Medicine in the first affiliated hospital of Guangzhou Medical University, Xuzhou maternity & child health hospital, Liwan hospital of traditional Chinese medicine, and Hexian memorial affiliated hospital of Southern Medical University if they meet the inclusion criteria and do not have any exclusion criteria. Eligible subjects will be approached and sign the consent form after detailed explanation of the study design and comprehensive counseling.

1.3 Screening visit Women will be screened in the morning after an overnight 12 hour fast. Detailed information about the study design will be given.

1.3.1 Sign informed consent Informed consent will be signed after detailed counseling. 1.3.2 Perform physical examination Perform complete physical examination including height, weight, hip, and waist measurement. Height and weight will be recorded to the nearest 0.1 cm and 0.1 kg respectively. Waist and hip circumference will be recorded to the nearest 1 cm. And assessment of hirsutism by FG, acne standard acne lesion counts, and pelvic exam.

1.3.3 Perform transvaginal ultrasound of ovaries Ovaries, including the ovarian size in three dimensions, the size of the largest ovarian follicle/cyst and size of every follicle with a mean diameter greater than 10 mm, and total antral follicle count (small follicles with mean diameter < 10 mm) of each ovary will be obtained through transvaginal ultrasound.

1.3.4 Check urine pregnancy test 1.3.5 Fasting blood samples to exclude other endocrine disorders Fasting (at least 4 h) blood samples will be taken to exclude any endocrine disorders:F-glucose, F-insulin, Hba1C (>7%), C-peptide, TSH (< 0.2 mIU/mL or >5.5 mIU/mL), T3 (<1.4 nmol/L or >2.2nmol/L), and free T4 (<10pmol/L or >23pmol/L).

1.3.6 Progestin withdrawal Prescribe progestin to induce withdrawal bleed, after eligibility is determined.

1.4 Baseline visit After screening visit, if a woman fulfills inclusion criteria and has signed the informed consent she will be assigned to the baseline visit. Baseline visit takes place day 2 - 5 of a spontaneous period or after a withdrawal bleeding after an overnight fast.

1.4.1 Laboratory Examination Collect 20ml of blood, and 10ml of blood will be for the following tests. The remaining 10ml of blood will be stored for determination of DNA and sphingolipid later.

1. Circulating sex steroids: Fasting serum levels of follicle-stimulating hormone (FSH), luteinizing hormone (LH), estrogen (E2), prolactin (PRL) and T, sex hormone binding globulin (SHBG), and dehydroepiandrosterone sulfate (DHEAS).
2. Lipid profile: Triglycerides (TG), total cholesterol (TC), high density lipoprotein (HDL-C), low density lipoprotein (LDL-C), apolipoprotein A1 (Apoa1), apolipoprotein B (ApoB), BRT, Renal, and Liver Profile.
3. Glucose homeostasis: The oral glucose tolerance test (OGTT) with 75 g glucose. Blood samples will be obtained to measure plasma glucose, serum insulin and C-peptide at 0, 60, and 120 min during the OGTT.

1.4.2 Complete questionnaires Quality of life will be assessed by the short form 36(SF-36), the Chinese Quality of Life (ChiQOL), sleeping questionnaires, international physical activity questionnaire (IPAQ) and the Polycystic Ovary Syndrome Questionnaire (PCOS-QOL). Investigators will also assess symptoms of anxiety and depression by the Zung SAS and Zung SDS questionnaires. And complete the quantization table of traditional Chinese medicine (TCM) syndromes about PCOS.

1.4.3 Assess TCM syndromes of patients Syndrome differentiation (Bian Zheng) in TCM is the comprehensive analysis of clinical information gained by the four main diagnostic TCM procedures: observation, listening, questioning, and pulse analysis, and it is used to guide the choice of treatment either by acupuncture and/or TCM herbal formulae. In PCOS, patients are empirically differentiated to be four categories: 1) phlegm-dampness syndrome, 2) blood stasis syndrome, 3) phlegm, and 4) blood stasis.

2. Intervention arms 2.1 Information to all study subjects All participants will be advised about the importance of regular physical exercise and a balanced diet by a trained dietician. Importantly, they will be instructed not to change their exercise or diet habits during the entire study period.

True acupuncture or, sham acupuncture and metformin/placebo will be started 2 days after the baseline visit including OGTT. All subjects will be asked to use a barrier method for contraception. True and sham acupuncture treatment will be given three times per week. Each treatment session lasts for 30 minutes and can be separated by an interval of 1-3 days, with a maximum of 90 treatment sessions during 4 month. After the third treatment, all patients fill in the expectation and credibility questionnaire. Metformin or placebo will be given at 0.5g/times, 3 times one day and for 4 month.

2.1.1 True acupuncture protocol The rationale of acupuncture protocols is based on Western Medical theories and the study protocol follows the CONSORT and STRICTA recommendations.Investigators will use fixed acupuncture protocols. The acupuncture protocol of this RCT follows the protocol in the following studies: ClinicalTrial.gov NCT01457209 and NCT02026323.

Disposable, single-use, sterilized needles made of stainless steel, 0.25 x 30 mm and 0.30 x 40/50 mm (Hwoto, Suzhou Medical Appliance Fact. 215005 Suzhou, China) will be inserted to a depth of 15-35 mm in segmental acupuncture points located in abdominal and leg muscles with innervations corresponding to the ovaries. Two sets of acupuncture points will be alternated every second treatment. The first set consists of conception vessel (CV) 4, CV 12, and stomach (ST) 29 bilaterally and in the muscles above the knee, ST 34, and ST 32 bilaterally and below the knee, spleen (SP) 6 and ST 36. Needles will also be placed in extra segmental acupuncture points that do not innervate the ovaries large intestine (LI) 4 bilaterally. In total 14 needles will be placed and all will be stimulated manually by rotating the needle to evoke needle sensation (de qi) once when inserted. The following points will be connected to an electrical stimulator (Export Abteilung, Schwa-Medico GmbH,Wetzlarer Str. 41-43;35630 Ehringshausen): CV 4 to CV 12, ST 29 bilateral, ST34 to ST 32 bilateral. Stimulation are given as low-frequency EA of 2Hz, 0.3 ms pulse length and with an intensity adjusted to produce local muscle contractions without pain or discomfort. Needles not connected to the electrical stimulator will be manually stimulated to evoke needle sensation every 10 min, in total 4 times. The second set consists of 14 needles placed in segmental abdominal points and stimulated electrically: ST 27 bilaterally, CV6 connected to CV10; and leg points: SP10 connected to a non-acupuncture point located 6 cun proximal of patellas medial border (electrical stimulation), and SP 6 and liver (LR) 3 bilaterally (manual stimulation). Extra segmental points are pericardium (PC) 6 bilaterally (manual stimulation).

2.1.2 Needle insertion technique Needle insertion should be gentle. Tighten the skin by pressing around the area of needle insertion and gently insert the needle.

2.1.3 Needles and stimulation Needle size: 0.25 x 30 mm or 0.30 x 40 or 0.30 x 50 mm. Select needle length with respect to the patients'BMI: 0.25 x 30 mm needles in women with normal BMI; 0.30 x 40 mm needles in overweight women and 0.30 x 50 or 75 mm needles in obese women. Depth of insertion may vary from patients to patients. Needles are placed with a depth deep enough to reach muscle/fibrous tissue. When needle are inserted, stimulate the needle gently until de qi (needle sensation reflecting activation of sensory afferents). As soon as de qi has been reached, make sure that the needle does not hurt or cause any pain and discomfort. Manual stimulation of needles that is not attached to an electrical stimulator (see below) are stimulated when inserted, after 10 minutes, 20 minutes and immediately before they are removed after 30 minutes.

Attach the electrodes according to the protocol. Turn on the stimulator (program 10) and increase the intensity. The intensity will be as high as possible without pain or discomfort. The stimulation amplitude/intensity will be adjusted after 10 and 20 minutes at the same time as when needle stimulated manually are manipulated. After 30 minutes the stimulator is turned off, electrodes disconnected and needles taken out.

2.1.4 Sham acupuncture protocol Disposable, single-use, sterilized needles made of stainless steel, 0.20 x 20 mm (Hwoto, Suzhou Medical Appliance Fact.215005 Suzhou, China) will be inserted superficially to a depth of <5 mm, one in each shoulder and on in each upper arm at non-acupuncture points. Placement of needles is unlikely to affect ovulation and IR in women with PCOS. Electrodes will be attached to the needles and the stimulator will be turned on at an intensity of zero (no active current) in order to mimic EA in the acupuncture protocol. No manual stimulation of the needles will be performed. An intended adjustment of the intensity after 10 minutes, 20 minutes and again after 30 minutes when stimulator is turned off and needles removed.

2.1.5 True and sham acupuncture treatment

1. Time of the day and acupuncturist name when the patient receives acupuncture will be recorded.
2. The intensity of stimulation (mA) is noted. It may vary between different electrodes. Note the range e.g. 1.2 - 3.0 mA.
3. Note any other events that may affect the treatment (positive or negative).
4. Note concomitant medications.
5. Collect menstrual logs at the end of every cycle. 2.2 Metformin and placebo Metformin (Kombiglyze XR) and placebo metformin will be packed and tested by a commercial pharmacy supply company (Squibb Company, Shanghai, China) specifically for this study. Metformin or placebo will be started 2 days after baseline visit including OGTT. Subjects will take 0.5 g/times, 3 times one day for up to 6 cycles.

2.3 Monitoring and examination during the treatment Physical examination will be performed monthly. Every menstruation should be recorded, including the date, volume and duration of menstruation during the entire study and follow-up. The condition of physical exercise and diet will be recorded for every cycle. OGTT will be repeated in the third month during the treatment.

2.4 End of treatment visit

During the end of treatment visit will all baseline measures be repeated as listed below:

1. Perform physical examination, including vital signs, height, weight, hip and waist measurements as well as repeating hirsutism and acne assessments after the end of treatment or pregnancy.
2. Repeat the serum levels of sex hormone steroids and metabolic profile.
3. Repeat transvaginal ultrasound of ovarian morphology.
4. Repeat OGTT.
5. Collect 20ml blood, and distributed store 10ml blood after serum separation. Other 10ml blood is for determination of DNA and sphingolipid.
6. Repeat QOL, sleeping, IPAQ anxiety/depression questionnaires, and the quantization table of TCM.
7. Collect menstrual logs.
8. Record adverse events and concomitant medications.
9. Answer the two questions about acupuncture treatment. 2.5 Follow-up visit Baseline and end of treatment visit will be repeated 3 months after last treatment (see point 1-8 under End of treatment visit). All the participants will be followed up with visiting the acupuncturists monthly for 3 month. The condition of physical exercise and diet will be record every month.

2.6 Safety analysis Adverse events will be categorized and percentage of patients experiencing adverse events and serious adverse events during the treatment period and follow up period will be documented. Chi-square tests will be performed to examine differences in the proportion of total and categories of adverse events.

2.7 Statistics One sample of the Kolmogorov-Smirnov test will be used to test the normal distribution of continuous variables. Continuous variables will be presented as means ± standard deviations if they are normally distributed or as medians with interquartile ranges if they are not normally distributed. Statistical comparison will be carried out according to the intention to treat by Student's t-test, Mann-Whitney U-test, and Wilcoxon signed ranks test for continuous variables and by χ2 tests for categorical variables where appropriate. All statistical analyses of the data will be performed using the SPSS program version 21.0 (SPSS Inc., Chicago, IL, USA), and a P-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese women aged from 18 to 40 years.
2. BMI ≥18.5kg/m2.
3. Confirmed diagnosis of PCOS according to modified Rotterdam criteria in 2003 including at least two of the following three features: ①Oligo-(an intermenstrual interval >35 days or <8 cycles in the past year), amenorrhea (an intermenstrual interval>90 days) and/or; ② polycystic ovarian morphology, i.e. presence of >12 antral follicles (≤ 9mm) and/or ovarian volume >10 ml on transvaginal scanning and/or; ③clinical and/or biochemical hyperandrogenism. Clinical hyperandrogenism in China Mainland is defined as a Ferriman-Gallwey (FG) score ≥5 ; biochemical hyperandrogenism is total testosterone (T) > 2.6 nmol/l and free testosterone ≥6.0 pg/ml.
4. Presence of IR as defined by the homeostatic model assessment (HOMA-IR: [fasting insulin (μU/mL) × fasting glucose (mmol/L)] / 22.5). A value ≥ 2.14 will be considered to be indicative of IR.
5. No immediate fertility wish and willingness to use barrier methods to contraception for one year.
6. Willingness to sign the consent form.

Exclusion Criteria:

1. Exclusion of other endocrine disorders:

   ① Uncorrected thyroid disease (defined as TSH < 0.2 mIU/mL or >5.5 mIU/mL). A normal level within the last year is adequate for entry.

   ② Poorly controlled of Type I or Type II diabetes (defined as a HbA1c level > 7.0%), or patients receiving antidiabetic medications such as insulin, thiazolidinediones, acarbose, or sulfonylureas likely to confound the effects of study medication; Patients currently receiving metformin XR (extended release) for a diagnosis of Type I or Type II diabetes or for PCOS are alsoexcluded.
   * Cushing's syndrome (define as an archetype of MetS. High glucocorticoid levels lead to muscle, liver and adipocyte insulin resistance. 17-OHCS>55umol/24h or UFC>304nmol/24h) ④ Congenital adrenal hyperplasia (define as patients with known 21-hydroxylase deficiency or other enzyme deficiency leading to the phenotype of congenital adrenal hyperplasia. 17-OHP>10 ng/ml in ACTH 1-24 h excited test (after 60 min)) ⑤ Suspected androgen secreting adrenal or ovarian tumor.
2. Use of hormonal or other medication including Chinese Herbal prescriptions which may affect the outcome the last 2 months.
3. Receiving acupuncture in the past 2 months.
4. Within 6 weeks pregnancy.
5. Post-abortion or postpartum within the past 6 weeks.
6. Breastfeeding within the last 4 months.
7. Not willing to give written consent to the study.
8. Having a bariatric surgery procedure within the past 12 months or being in a period of acute weight loss.
9. Additional exclusion criteria including:

   * Patients on oral contraceptives, depot progestins, or hormonal implants (including Implanon). A two month washout period will be required prior to screening for patients on these agents. Longer washouts may be necessary for certain depot contraceptive forms or implants, especially where the implants are still in place. A one-month washout will be required for patients on oral cyclic progestins.

     * Heart disease ③ Patients with a history of, or suspected cervical carcinoma, endometrial carcinoma, or breast carcinoma.

       * Patients enrolled into other studies that require medications. ⑤ Patients taking longer than a one month break during the protocol should not be enrolled.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 342 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Changes of HOMA-IR | Change from Baseline Systolic Blood Pressure at 4 months and 7 months

SECONDARY OUTCOMES:
HOMA-B | 4 months and 7 months
AUCglu | 4 months and 7 months
Menstrual frequency | 4 months and 7 months
Body composition（a composite） | 4 months and 7 months
  Weight, BMI, waist-to-hip circumference, FG and acne lesion counts
Metabolic profile（a composite） | 4 months and 7 months
  Glucose and insulin concentrations, C-peptide, HbA1c, TC, TG, HDL-C and LDL-C, ApoA1 and ApoB.
Hormonal profile（a composite） | 4 months and 7 months
  FSH, LH, T, SHBG and DHEAS
Questionnaires（a composite） | 4 months and 7 months
  SF-36, ChiQOL, sleeping questionnaires, IPAQ, PCOS-QOL, Zung SAS, Zung SDS questionnaires and the quantization table of TCM syndromes about PCOS
Side effect profile | 4 months and 7 months
Expectation and credibility of treatment（questionnaire, 6 questions，4grades，0-24scores) | 1 week and 4 months
AUCins | 4 months and 7 months
Ovulation rate | 4 months and 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Ma, Study Chair — The First Affiliated Hospital of Guangzhou Medical University; Juan Li, PhD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Maohua Lai, PhD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Hua Liu, Master, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Wanting Wu, Master, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Ernest HY NG, PhD, Principal Investigator — The University of Hong Kong; Elisabet Stener-Victorin, PhD, Study Director — Karolinska Institutet
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lakkakula BV, Thangavelu M, Godla UR. Genetic variants associated with insulin signaling and glucose homeostasis in the pathogenesis of insulin resistance in polycystic ovary syndrome: a systematic review. J Assist Reprod Genet. 2013 Jul;30(7):883-95. doi: 10.1007/s10815-013-0030-1. Epub 2013 Jun 22. PMID 23794114
- [Background] Nestler JE. Role of hyperinsulinemia in the pathogenesis of the polycystic ovary syndrome, and its clinical implications. Semin Reprod Endocrinol. 1997 May;15(2):111-22. doi: 10.1055/s-2007-1016294. PMID 9165656
- [Background] Farrell K, Antoni MH. Insulin resistance, obesity, inflammation, and depression in polycystic ovary syndrome: biobehavioral mechanisms and interventions. Fertil Steril. 2010 Oct;94(5):1565-74. doi: 10.1016/j.fertnstert.2010.03.081. Epub 2010 May 14. PMID 20471009
- [Background] Bhathena RK. Insulin resistance and the long-term consequences of polycystic ovary syndrome. J Obstet Gynaecol. 2011;31(2):105-10. doi: 10.3109/01443615.2010.539722. PMID 21281021
- [Background] Hernandez-Valencia M, Hernandez-Rosas M, Zarate A. [Care of insulin resistance in polycystic ovary syndrome]. Ginecol Obstet Mex. 2010 Nov;78(11):612-6. Spanish. PMID 21298999
- [Background] Franks S. When should an insulin sensitizing agent be used in the treatment of polycystic ovary syndrome? Clin Endocrinol (Oxf). 2011 Feb;74(2):148-51. doi: 10.1111/j.1365-2265.2010.03934.x. PMID 21121941
- [Background] Pauli JM, Raja-Khan N, Wu X, Legro RS. Current perspectives of insulin resistance and polycystic ovary syndrome. Diabet Med. 2011 Dec;28(12):1445-54. doi: 10.1111/j.1464-5491.2011.03460.x. PMID 21950959
- [Background] Zhou G, Myers R, Li Y, Chen Y, Shen X, Fenyk-Melody J, Wu M, Ventre J, Doebber T, Fujii N, Musi N, Hirshman MF, Goodyear LJ, Moller DE. Role of AMP-activated protein kinase in mechanism of metformin action. J Clin Invest. 2001 Oct;108(8):1167-74. doi: 10.1172/JCI13505. PMID 11602624
- [Background] Hwang KR, Choi YM, Kim JJ, Chae SJ, Park KE, Jeon HW, Ku SY, Kim SH, Kim JG, Moon SY. Effects of insulin-sensitizing agents and insulin resistance in women with polycystic ovary syndrome. Clin Exp Reprod Med. 2013 Jun;40(2):100-5. doi: 10.5653/cerm.2013.40.2.100. Epub 2013 Jun 30. PMID 23875167
- [Background] Legro RS, Arslanian SA, Ehrmann DA, Hoeger KM, Murad MH, Pasquali R, Welt CK; Endocrine Society. Diagnosis and treatment of polycystic ovary syndrome: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2013 Dec;98(12):4565-92. doi: 10.1210/jc.2013-2350. Epub 2013 Oct 22. PMID 24151290
- [Background] Chang CT, Chen YC, Fang JT, Huang CC. Metformin-associated lactic acidosis: case reports and literature review. J Nephrol. 2002 Jul-Aug;15(4):398-402. PMID 12243370
- [Background] Triggle CR, Ding H. Cardiovascular impact of drugs used in the treatment of diabetes. Ther Adv Chronic Dis. 2014 Nov;5(6):245-68. doi: 10.1177/2040622314546125. PMID 25364492
- [Background] Dunaif A. Drug insight: insulin-sensitizing drugs in the treatment of polycystic ovary syndrome--a reappraisal. Nat Clin Pract Endocrinol Metab. 2008 May;4(5):272-83. doi: 10.1038/ncpendmet0787. Epub 2008 Mar 25. PMID 18364705
- [Background] Graham DJ, Ouellet-Hellstrom R, MaCurdy TE, Ali F, Sholley C, Worrall C, Kelman JA. Risk of acute myocardial infarction, stroke, heart failure, and death in elderly Medicare patients treated with rosiglitazone or pioglitazone. JAMA. 2010 Jul 28;304(4):411-8. doi: 10.1001/jama.2010.920. Epub 2010 Jun 28. PMID 20584880
- [Background] Mamtani R, Haynes K, Bilker WB, Vaughn DJ, Strom BL, Glanz K, Lewis JD. Association between longer therapy with thiazolidinediones and risk of bladder cancer: a cohort study. J Natl Cancer Inst. 2012 Sep 19;104(18):1411-21. doi: 10.1093/jnci/djs328. Epub 2012 Aug 9. PMID 22878886
- [Background] Betteridge DJ. Thiazolidinediones and fracture risk in patients with Type 2 diabetes. Diabet Med. 2011 Jul;28(7):759-71. doi: 10.1111/j.1464-5491.2010.03187.x. PMID 21672000
- [Background] Witt CM, Pach D, Brinkhaus B, Wruck K, Tag B, Mank S, Willich SN. Safety of acupuncture: results of a prospective observational study with 229,230 patients and introduction of a medical information and consent form. Forsch Komplementmed. 2009 Apr;16(2):91-7. doi: 10.1159/000209315. Epub 2009 Apr 9. PMID 19420954
- [Background] Stener-Victorin E, Jedel E, Janson PO, Sverrisdottir YB. Low-frequency electroacupuncture and physical exercise decrease high muscle sympathetic nerve activity in polycystic ovary syndrome. Am J Physiol Regul Integr Comp Physiol. 2009 Aug;297(2):R387-95. doi: 10.1152/ajpregu.00197.2009. Epub 2009 Jun 3. PMID 19494176
- [Background] Manni L, Rocco ML, Barbaro Paparo S, Guaragna M. Electroacupucture and nerve growth factor: potential clinical applications. Arch Ital Biol. 2011 Jun;149(2):247-55. doi: 10.4449/aib.v149i2.1365. PMID 21701996
- [Background] Liang F, Koya D. Acupuncture: is it effective for treatment of insulin resistance? Diabetes Obes Metab. 2010 Jul;12(7):555-69. doi: 10.1111/j.1463-1326.2009.01192.x. PMID 20590731
- [Background] Johansson J, Manneras-Holm L, Shao R, Olsson A, Lonn M, Billig H, Stener-Victorin E. Electrical vs manual acupuncture stimulation in a rat model of polycystic ovary syndrome: different effects on muscle and fat tissue insulin signaling. PLoS One. 2013;8(1):e54357. doi: 10.1371/journal.pone.0054357. Epub 2013 Jan 18. PMID 23349861
- [Background] Benrick A, Maliqueo M, Johansson J, Sun M, Wu X, Manneras-Holm L, Stener-Victorin E. Enhanced insulin sensitivity and acute regulation of metabolic genes and signaling pathways after a single electrical or manual acupuncture session in female insulin-resistant rats. Acta Diabetol. 2014 Dec;51(6):963-72. doi: 10.1007/s00592-014-0645-4. Epub 2014 Sep 14. PMID 25218925
- [Background] Zhao X, Ni R, Li L, Mo Y, Huang J, Huang M, Azziz R, Yang D. Defining hirsutism in Chinese women: a cross-sectional study. Fertil Steril. 2011 Sep;96(3):792-6. doi: 10.1016/j.fertnstert.2011.06.040. Epub 2011 Jul 18. PMID 21762890
- [Background] Ni RM, Mo Y, Chen X, Zhong J, Liu W, Yang D. Low prevalence of the metabolic syndrome but high occurrence of various metabolic disorders in Chinese women with polycystic ovary syndrome. Eur J Endocrinol. 2009 Sep;161(3):411-8. doi: 10.1530/EJE-09-0298. Epub 2009 Jun 19. PMID 19542239
- [Background] Chen X, Yang D, Li L, Feng S, Wang L. Abnormal glucose tolerance in Chinese women with polycystic ovary syndrome. Hum Reprod. 2006 Aug;21(8):2027-32. doi: 10.1093/humrep/del142. Epub 2006 May 9. PMID 16684838
- [Background] McHorney CA, Ware JE Jr, Raczek AE. The MOS 36-Item Short-Form Health Survey (SF-36): II. Psychometric and clinical tests of validity in measuring physical and mental health constructs. Med Care. 1993 Mar;31(3):247-63. doi: 10.1097/00005650-199303000-00006. PMID 8450681
- [Background] Cronin L, Guyatt G, Griffith L, Wong E, Azziz R, Futterweit W, Cook D, Dunaif A. Development of a health-related quality-of-life questionnaire (PCOSQ) for women with polycystic ovary syndrome (PCOS). J Clin Endocrinol Metab. 1998 Jun;83(6):1976-87. doi: 10.1210/jcem.83.6.4990. PMID 9626128
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Leung KF, Liu FB, Zhao L, Fang JQ, Chan K, Lin LZ. Development and validation of the Chinese Quality of Life Instrument. Health Qual Life Outcomes. 2005 Apr 16;3:26. doi: 10.1186/1477-7525-3-26. PMID 15833138
- [Background] Jiang M, Lu C, Zhang C, Yang J, Tan Y, Lu A, Chan K. Syndrome differentiation in modern research of traditional Chinese medicine. J Ethnopharmacol. 2012 Apr 10;140(3):634-42. doi: 10.1016/j.jep.2012.01.033. Epub 2012 Feb 1. PMID 22322251
- [Background] Moher D, Schulz KF, Altman D; CONSORT Group. The CONSORT Statement: revised recommendations for improving the quality of reports of parallel-group randomized trials 2001. Explore (NY). 2005 Jan;1(1):40-5. doi: 10.1016/j.explore.2004.11.001. PMID 16791967
- [Background] MacPherson H, Altman DG, Hammerschlag R, Youping L, Taixiang W, White A, Moher D; STRICTA Revision Group. Revised STandards for Reporting Interventions in Clinical Trials of Acupuncture (STRICTA): extending the CONSORT statement. PLoS Med. 2010 Jun 8;7(6):e1000261. doi: 10.1371/journal.pmed.1000261. PMID 20543992
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Iwata M, Maeda S, Kamura Y, Takano A, Kato H, Murakami S, Higuchi K, Takahashi A, Fujita H, Hara K, Kadowaki T, Tobe K. Genetic risk score constructed using 14 susceptibility alleles for type 2 diabetes is associated with the early onset of diabetes and may predict the future requirement of insulin injections among Japanese individuals. Diabetes Care. 2012 Aug;35(8):1763-70. doi: 10.2337/dc11-2006. Epub 2012 Jun 11. PMID 22688542
- [Background] Kahn SE, Prigeon RL, McCulloch DK, Boyko EJ, Bergman RN, Schwartz MW, Neifing JL, Ward WK, Beard JC, Palmer JP, et al. Quantification of the relationship between insulin sensitivity and beta-cell function in human subjects. Evidence for a hyperbolic function. Diabetes. 1993 Nov;42(11):1663-72. doi: 10.2337/diab.42.11.1663. PMID 8405710
- [Background] Zheng Y, Stener-Victorin E, Ng EH, Li J, Wu X, Ma H. How does acupuncture affect insulin sensitivity in women with polycystic ovary syndrome and insulin resistance? Study protocol of a prospective pilot study. BMJ Open. 2015 May 3;5(4):e007757. doi: 10.1136/bmjopen-2015-007757. PMID 25941189
- [Derived] Wen Q, Hu M, Lai M, Li J, Hu Z, Quan K, Liu J, Liu H, Meng Y, Wang S, Wen X, Yu C, Li S, Huang S, Zheng Y, Lin H, Liang X, Lu L, Mai Z, Zhang C, Wu T, Ng EHY, Stener-Victorin E, Ma H. Effect of acupuncture and metformin on insulin sensitivity in women with polycystic ovary syndrome and insulin resistance: a three-armed randomized controlled trial. Hum Reprod. 2022 Mar 1;37(3):542-552. doi: 10.1093/humrep/deab272. PMID 34907435
- [Derived] Li J, Ng EH, Stener-Victorin E, Hu Z, Shao X, Wang H, Li M, Lai M, Xie C, Su N, Yu C, Liu J, Wu T, Ma H. Acupuncture treatment for insulin sensitivity of women with polycystic ovary syndrome and insulin resistance: a study protocol for a randomized controlled trial. Trials. 2017 Mar 9;18(1):115. doi: 10.1186/s13063-017-1854-2. PMID 28274268